CLINICAL TRIAL: NCT05851521
Title: HERMES Study: A Randomized Clinical Trial To Evaluate Lower Urinary Tract Symptoms Differences Between Indwelling Catheter And Temporary Prostatic Stent In Patients Undergoing Minimally Invasive Procedures For The Treatment Of Localized Prostate Cancer Or Benign Prostatic Hyperplasia
Brief Title: To Evaluate LUTS and Complications Between Indwelling Catheter and Temporary Prostatic Stent in Patients Undergoing Minimally Invasive Procedures for the Treatment of Localized Prostate Cancer or Benign Prostatic Hyperplasia (HERMES)
Acronym: HERMES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lyx Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HERMES01
Record Dates: First submitted 2023-03-22; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Lower Urinary Tract Symptoms; Prostatic Hyperplasia; Prostatic Cancer; Urinary Retention
Keywords: Temporary prostatic stent; Indwelling catheter; Cryotherapy; Prostate cancer; Benign prostatic hyperplasia; Rezum; EchoLaser
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Prostatic Hyperplasia; Prostatic Neoplasms; Urinary Retention | interventions — Catheters, Indwelling

STUDY DESIGN:
Intervention Model Description: Prospective randomized clinical trial divided in 3 cohorts: HERMES_CRYO (cryotherapy for targeted therapy of localized prostate cancer), HERMES_REZUM [water vapor energy ablation for the treatment of benign prostatic hyperplasia (BPH)], and HERMES_LASER [ELESTA ECHOLASER® for the treatment of benign prostatic hyperplasia (BPH)].
  In each cohort, two arms will be compared: temporary prostatic stent vs indwelling catheter with a 1:1 randomization ratio.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Temporary prostatic stent (Exime®) (Experimental): Post-operative placement of temporary prostatic stent (EXIME)
  Interventions: Device: Temporary prostatic stent (Exime®)
- Indwelling catheter (Active Comparator): Post-operative placement of indwelling catheter
  Interventions: Device: Indwelling catheter

INTERVENTIONS:
Device: Temporary prostatic stent (Exime®) — Placement of temporary prostatic stent (Exime®) following the procedure described in the product information
  Arms: Temporary prostatic stent (Exime®)
Device: Indwelling catheter — Placement of indwelling catheter
  Arms: Indwelling catheter

SUMMARY:
The goal of this single-centre prospective randomized clinical trial is to compare the post-operative use of temporary prostatic stent (Group 1) vs indwelling catheter (Group 2) in patients undergoing cryotherapy for targeted therapy of localized prostate cancer, transurethral water vapor energy ablation (REZUM) or transperineal laser ablation of the prostate with EchoLaser™ system for the treatment of benign prostatic hyperplasia (BPH)

The main questions are:

* Difference in quality of life, Lower Urinary Tract Symptoms (scored with IPSS, International Prostate Symptom Score), urinary continence symptoms (scored with International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form, ICIQ-UI-SF) and patient satisfaction between indwelling catheter and temporary prostatic stent (Exime®) score with a non-validated questionnaire (Stent/catheter-related urinary symptoms questionnaire)
* Difference in side effects and complications between indwelling catheter and temporary prostatic stent (Exime®)

A total 120 of patients will be enrolled (Group 1: 60; Group 2: 60) with a 1:1 randomization ratio. The follow-up duration will be 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent prior to enrollment (if applicable).
* Subjects must meet all inclusion criteria to be eligible for study enrollment.
* Men between 18 and 85 years old.
* Undergo focal therapy for prostate cancer, water vapour energy ablation Rezum® or EchoLaser®.
* Willing to be seen by the investigator and answer questions and fill out questionnaires up to a month after surgery.

Exclusion Criteria:

* Urethral stricture <22F.
* Gross haematuria
* Prostate volume > 80cc
* Prostate craniocaudal length > 6cm
* Patients with long-term urinary catheters or other urinary drainage systems
* Lack of commitment on the part of the patient to attend the follow-up as required.

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Device-related quality of life | 1 week
  Evaluation of impact on patient quality of life associated with the urinary device will be based on the sixth question (Q6) of a non validated questionnaire (Stent/catheter-related urinary symptoms questionnaire), defined as:
  Q6: "How much has the bladder catheter/Exime affected your quality of life?" Quantitative answer, ranging from 0 to 10. Being zero, not affected; and being ten, very affected

SECONDARY OUTCOMES:
Device-related urinary side effects | 1 week
  Evaluation will be based on the first five questions (Q1 - Q5) of a non validated questionnaire with quantitative answers ranging from 0 to 10, defined as:
  Q1:How much urine leakage have you had while carrying the bladder catheter or the Exime® device? (0: none -> 10 a lot of leakage = need to use several diapers) Q2. How much pain, discomfort or spasms have you had in relation to the catheter/Exime®? (0: none -> 10: a lot of pain = need for prescribed analgesia) Q3. How much bleeding have you had with urine while wearing the catheter/Exime®? (0: none -> 10: a lot of bleeding = need for change of clothing) Q4. How much has the urine been different? (darker than usual, worse odor, or sediment)? (0: nothing -> 10: very strong odor, very dark urine, presence of lumps) Q5. Have you had any problems in handling the catheter? (0: no problems at all -> 10: many problems)
Device-related patient satisfaction | 1 week
  Evaluation of satisfaction of patients associated with the device will be based on the seventh question (Q7) of a non validated questionnaire (Stent/catheter-related urinary symptoms questionnaire), defined as:
  Q7. What is your degree of satisfaction while wearing the catheter/Exime®? Quantitative answer, ranging from 0 to 10. Being zero, not satisfied at all; and being ten, completely satisfied
Device-related Lower Urinary Tract Symptoms (LUTS) | From device-placement to 6 months after treatment
  Evaluation of impact of the device on LUTS will be based on a validated questionnaire administered before the device-placement, at device-removal, at 4 weeks and finally at 6 months after treatment:
  - International Prostate Symptom Score (IPSS), min 0 - max 35 points, in which higher values are associated with worsening urinary symptoms
Occurence of perioperative events (< or = 24h after treatment) | 1 post-operative day
  Evaluation of perioperative events (< or = 24h after treatment) defined as complications (classified according to the Clavien - Dindo scale), presence of haematuria, pain (based on visual analogue pain score), occurence of acute urinary retention or need to perform urinary catheter bladder washout.
Occurrence of postoperative events (>24h-1week) | 1 week
  Evaluation of postoperative events (>24h-1week) defined as acute urinary retention or need to perform urinary catheter bladder washout, need to change urinary catheter or presence of urinary tract infection (presence of fever or need to change antibiotic therapy) and others complications (classified according to the Clavien - Dindo scale)
Overall satisfaction outcomes | 4 week
  Evaluation of overall satisfaction will be based on the question "How satisfied are you overall with the treatment you have received? (Quantitative answer, ranging from 0 to 10. Being zero, not satisfied at all; and being ten, completely satisfied) administered at 4 week post-treatment.
Urine flow rate | From device-placement to 6 months after treatment
  Maximal flow rate [Q max (ml/s)] will be evaluated performing a uroflowmetry at baseline, at week 4, and finally at 6 months after treatment.
Device-related continence symptoms | From device-placement to 6 months after treatment
  Evaluation of impact of the device on continence symptoms will be based on a validated questionnaire administered before the device-placement, at device-removal, at 4 weeks and finally at 6 months after treatment:
  - International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI-SF): min 0 - max 21 points, the higher the score, the more severe is the urinary incontinence, but there is no normal score.

CONTACTS AND LOCATIONS:
Overall Officials: Juan I Martinez-Salamanca, MD PhD FEBU FACS FEBSM, Principal Investigator — Lyx Institute Urología
Locations (1):
- Juan Ignacio Martinez-Salamanca, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Drinka PJ. Complications of chronic indwelling urinary catheters. J Am Med Dir Assoc. 2006 Jul;7(6):388-92. doi: 10.1016/j.jamda.2006.01.020. Epub 2006 Mar 23. PMID 16843240
- [Result] Toughill E. Indwelling urinary catheters: common mechanical and pathogenic problems. Am J Nurs. 2005 May;105(5):35-7. doi: 10.1097/00000446-200505000-00025. No abstract available. PMID 15867530
- [Result] Parsons JK. Benign Prostatic Hyperplasia and Male Lower Urinary Tract Symptoms: Epidemiology and Risk Factors. Curr Bladder Dysfunct Rep. 2010 Dec;5(4):212-218. doi: 10.1007/s11884-010-0067-2. Epub 2010 Sep 7. PMID 21475707
- [Result] Patelli G, Ranieri A, Paganelli A, Mauri G, Pacella CM. Transperineal Laser Ablation for Percutaneous Treatment of Benign Prostatic Hyperplasia: A Feasibility Study. Cardiovasc Intervent Radiol. 2017 Sep;40(9):1440-1446. doi: 10.1007/s00270-017-1662-9. Epub 2017 May 4. PMID 28474112
- [Result] McVary KT, Rogers T, Roehrborn CG. Rezum Water Vapor Thermal Therapy for Lower Urinary Tract Symptoms Associated With Benign Prostatic Hyperplasia: 4-Year Results From Randomized Controlled Study. Urology. 2019 Apr;126:171-179. doi: 10.1016/j.urology.2018.12.041. Epub 2019 Jan 21. PMID 30677455
- [Result] Westwood J, Geraghty R, Jones P, Rai BP, Somani BK. Rezum: a new transurethral water vapour therapy for benign prostatic hyperplasia. Ther Adv Urol. 2018 Aug 12;10(11):327-333. doi: 10.1177/1756287218793084. eCollection 2018 Nov. PMID 30344644
- [Result] Fernandez-Guzman E, Asensio Matas A, Capape Poves V, Rioja Zuazu J, Garrido Abad P, Martinez-Salamanca JI, Quintana Franco LM, Justo-Quintas J, Romero-Otero J, Dominguez-Esteban M. Preliminary results of a national multicenter study on the treatment of LUTS secondary to benign prostatic hyperplasia using the Rezum(R) steam system. Actas Urol Esp (Engl Ed). 2022 Jun;46(5):310-316. doi: 10.1016/j.acuroe.2021.11.003. Epub 2022 May 12. English, Spanish. PMID 35570100
- [Result] Helo S, Holland B, McVary KT. Convective Radiofrequency Water Vapor Thermal Therapy with Rezum System. Curr Urol Rep. 2017 Oct;18(10):78. doi: 10.1007/s11934-017-0728-1. PMID 28780635
- [Result] Guelce D, Thomas D, Elterman D, Chughtai B. Recent advances in managing benign prostatic hyperplasia: The Rezum System. F1000Res. 2018 Dec 10;7:F1000 Faculty Rev-1916. doi: 10.12688/f1000research.15851.1. eCollection 2018. PMID 30631433
- [Result] Avery K, Donovan J, Peters TJ, Shaw C, Gotoh M, Abrams P. ICIQ: a brief and robust measure for evaluating the symptoms and impact of urinary incontinence. Neurourol Urodyn. 2004;23(4):322-30. doi: 10.1002/nau.20041. PMID 15227649
- [Result] Lebastchi AH, George AK, Polascik TJ, Coleman J, de la Rosette J, Turkbey B, Wood BJ, Gorin MA, Sidana A, Ghai S, Tay KJ, Ward JF, Sanchez-Salas R, Muller BG, Malavaud B, Mozer P, Crouzet S, Choyke PL, Ukimura O, Rastinehad AR, Pinto PA. Standardized Nomenclature and Surveillance Methodologies After Focal Therapy and Partial Gland Ablation for Localized Prostate Cancer: An International Multidisciplinary Consensus. Eur Urol. 2020 Sep;78(3):371-378. doi: 10.1016/j.eururo.2020.05.018. Epub 2020 Jun 10. PMID 32532513
- [Result] Shah TT, Peters M, Eldred-Evans D, Miah S, Yap T, Faure-Walker NA, Hosking-Jervis F, Thomas B, Dudderidge T, Hindley RG, McCracken S, Greene D, Nigam R, Valerio M, Minhas S, Winkler M, Arya M, Ahmed HU. Early-Medium-Term Outcomes of Primary Focal Cryotherapy to Treat Nonmetastatic Clinically Significant Prostate Cancer from a Prospective Multicentre Registry. Eur Urol. 2019 Jul;76(1):98-105. doi: 10.1016/j.eururo.2018.12.030. Epub 2019 Jan 9. PMID 30638633
- [Result] Eggener SE, Scardino PT, Carroll PR, Zelefsky MJ, Sartor O, Hricak H, Wheeler TM, Fine SW, Trachtenberg J, Rubin MA, Ohori M, Kuroiwa K, Rossignol M, Abenhaim L; International Task Force on Prostate Cancer and the Focal Lesion Paradigm. Focal therapy for localized prostate cancer: a critical appraisal of rationale and modalities. J Urol. 2007 Dec;178(6):2260-7. doi: 10.1016/j.juro.2007.08.072. Epub 2007 Oct 15. PMID 17936815